CLINICAL TRIAL: NCT05785429
Title: The Effect of Colchicine on Food-related Effort-based Decision Making in Brain and Behaviour in Overweight and Obesity: the FLAIR-i Study
Brief Title: The Effect of Colchicine on Food-related Effort-based Decision Making in Brain and Behaviour in Overweight and Obesity
Acronym: FLAIR-i
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Donders Centre for Cognitive Neuroimaging (Other)
Collaborators: Radboud University Medical Center (Other); HAN University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 3033002.01; 2021-004919-11 (EudraCT Number)
Record Dates: First submitted 2022-09-27; First posted 2023-03-27 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; Inflammation; fMRI; Motivation
MeSH Terms: conditions — Overweight; Obesity; Inflammation | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Experimental): One tablet of colchicine 0.5 mg per day
  Interventions: Drug: Colchicine 0.5 MG
- Placebo (Placebo Comparator): One tablet of microcrystalline cellulose per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 MG — Participant in the intervention group receive one tablet of 0.5mg colchicine per day for 12 weeks.
  Arms: Colchicine
Drug: Placebo — Participants in the intervention group receive one tablet of placebo per day for 12 weeks.
  Arms: Placebo

SUMMARY:
The main objective of the FLAIR-i study is to study the causal role of inflammation in affecting effort-based decision making in brain and behaviour in overweight and obesity, by comparing the effect of the anti-inflammatory agent colchicine vs. placebo.

DETAILED DESCRIPTION:
Obesity is a major health problem worldwide and is characterized by increases in low-grade, systemic inflammation. Outside the field of obesity, increases in inflammation have been related to loss of motivation and effortful behaviour, which can be objectively measured with effort-based decision making in brain and behaviour. Here, the investigators hypothesise that low-grade inflammation is causing altered striatal brain responses and effortless 'fast food' choices in overweight and obesity. The objective of this study is to study the causal role of inflammation in affecting effort-based decision making in brain and behaviour in overweight and obese participants, by comparing the effect of the anti-inflammatory agent colchicine vs. placebo. In addition, it will be investigated whether this primary objective translates to more ecologically valid measures/settings.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27 kg/m2
* Female sex
* Right-handed
* Age: 18-59 years
* Shoulder width of < 68 cm (to fit into the MRI scanner)
* Dutch speaking - Sufficient level to understand task instructions
* Low-grade inflammatory state, as measured by C-reactive protein (CRP) between 3.0 and 10.0 mg/L

Exclusion Criteria:

* Having been vaccinated by any type of vaccine in the 4 weeks preceding the first test session
* Having had an infection characterized by a fever, or diagnosed by a medical physician in the 4 weeks preceding the first test session
* Diagnosed with Diabetes Mellitus type I or II
* Gained or lost >2 points in BMI (kg/m2) over the last 6 months
* Followed an energy restricting diet during the last 2 months
* Having had bariatric surgery in the past 5 years
* Regular use of anti-inflammatory, anti-diabetic, weight-loss, and psychoactive medication
* Regular use of CYP3A4 inhibitors, P-glycoprotein inhibitors, statins, fibrates, ciclosporin, and digoxin, as a contraindication for colchicine
* Have renal impairment as evidenced by serum creatinine >150 μmol/l or eGFR <50mL/min/1.73m2, determined maximum 12 weeks before inclusion
* Have moderate to severe hepatic disease
* (History of) clinically significant psychiatric or neurological disorder
* (History of) clinically significant metabolic, cardiovascular, renal, liver, endocrinological, autoimmune or chronic inflammatory disease
* General medical conditions, such as sensorimotor handicaps, deafness, blindness or colour-blindness, as judged by the investigator
* Current or history of alcohol and/or drugs abuse (i.e. >14 units per week)
* Habitual smoking, i.e. one or more cigarettes per day
* Pregnant, lactating or wishing to become pregnant in the period between the screening and until 3 months after the last study visit
* Participation in another weight loss, lifestyle or anti-inflammatory intervention in the context of research at the time of inclusion or during the study
* Contraindications for MRI

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Change in effort valuation in brain and behaviour | Change between baseline and follow-up after 12 weeks
  Brain activity (BOLD signal during functional MRI) and behavioural weightings upon/of effort sensitivity, as measured by an effort-based decision making task.
Change in reward valuation in brain and behaviour | Change between baseline and follow-up after 12 weeks
  Brain activity (BOLD signal during functional MRI) and behavioural weightings upon/of reward sensitivity, as measured by an effort-based decision making task.

SECONDARY OUTCOMES:
Change effort/reward related food intake ratio | Change between baseline and follow-up after 12 weeks
  Intake of food items varying in effort and reward/calories, measured by a bogus food taste test.
Change in reward anticipation/reward consummation ratio in daily life | Change between baseline and follow-up after 12 weeks
  Reward anticipation and reward consummation scores in daily life as measured by the Experience Sampling Method

OTHER OUTCOMES:
C-reactive protein | Change between baseline and follow-up after 12 weeks
  High sensitive C-reactive protein measured in plasma
Inflammation profile (blood) | Change between baseline and follow-up after 12 weeks
  Assay-based profile of systemic inflammation measured in plasma stimulation, Olink Inflammatory profile
Brain myo-inositol levels | Change between baseline and follow-up after 12 weeks
  Brain myo-inositol levels reflecting neuroinflammation in ventral striatum and ACC, measured by magnetic resonance spectroscopy
Abdominal fat distribution | Change between baseline and follow-up after 12 weeks
  VAT(visceral adipose tissue)/SAT(subcutaneous adipose tissue) ratio based on abdominal MRI scan
(Resting state) functional connectivity networks | Change between baseline and follow-up after 12 weeks
  Measured by functional MRI

CONTACTS AND LOCATIONS:
Overall Officials: Esther Aarts, Prof.dr., Principal Investigator — Donders Centre for Cognitive Neuroimaging
Locations (1):
- Donders Centre for Cognitive Neuroimaging, Nijmegen, Netherlands